CLINICAL TRIAL: NCT06415539
Title: The Effect of Vestibular and Proprioceptive Exercise Practices on Hyperactivity Levels in Children With Autism Spectrum Disorder
Brief Title: The Effect of Exercise Practices on Hyperactivity Levels in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar10
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Classic physical therapy program will be applied
  Interventions: Other: classical physical therapy program
- exercise (Experimental): In addition to the classical physical therapy program, a treatment program including vestibular and proprioceptive exercise training will be applied.
  Interventions: Other: classical physical therapy program; Other: exercises

INTERVENTIONS:
Other: classical physical therapy program — Children in the control group, where classical physiotherapy and rehabilitation methods are applied, will continue their individual training programs with a physiotherapist for 40 minutes, 2 days a week, for 8 weeks.
Other: exercises — Children in this group will be given vestibular and proprioceptive exercise training in addition to the classical physiotherapy program. Skateboard, swing, hammock, bowl, ball, sensory pads, ball pool, slide, climbing bar, trampoline and balance board will be used as materials in vestibular and proprioceptive exercise training. In addition, at the end of the training sessions, parents will be informed about the application of exercise training to daily activities.
  Arms: exercise

SUMMARY:
The aim of this study is to examine the effect of vestibular and proprioceptive exercise practices on the hyperactivity level in children with autism spectrum disorder.

DETAILED DESCRIPTION:
The families of all children participating in the study will be informed and their written consent will be obtained. Vestibular and proprioceptive evaluation, hyperactivity evaluation and nystagmus evaluation will be applied to each child participating in the study twice, before and after treatment. Children will be divided into two groups: an exercise group and a control group, consisting of equal numbers of patients. A classical physical therapy program will be applied to both groups. In addition to the exercise group, a treatment program including vestibular and proprioceptive exercise training will be applied. The training program for both groups will be held in 40-minute sessions, 2 days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* children whose voluntary consent form is signed by their parents
* Children ages 6 to 10
* not using supplements
* not having undergone any surgical operation

Exclusion Criteria:

* children who have any obstacle to exercise
* They were determined as children who could not cooperate in the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Postrotary Nystagmus Assessment Test | 8 weeks
  The most common diagnostic assessment for vestibular function includes use of the postrotary nystagmus test17 and clinical observation. The postrotary nystagmus test is used to identify whether a child has a vestibular disability During the test, the subject is seated on a rotation disk, with his or her head fixed in a 30-degree angle forward, to ensure that the semicircular canals are horizontal.19 Next, the subject is rotated for ten clockwise or counterclockwise rotations, at 2 seconds per rotation. The subject is asked to gaze forward with both eyes, and the examiner observes the degree of nystagmus produced by the rotations.
Sensory Profile Test | 8 weeks
  Sensory Profile is a report-based questionnaire that is applied to measure the sensory processing abilities of children between the ages of 3-10 and to reveal the effects of the sensory processing process on the functional performance of children in their daily lives, and can determine children's sensory performances in detail. The survey can be applied to children with different types and degrees of disability. Mother, father or caregiver; That is, the evaluation is carried out by the people who are primarily responsible for the child's care by rating the 33 items in the survey according to their frequency. Items are scored as "always = 1, often = 2, sometimes = 3, rarely = 4, never = 5". Raw score totals for each section and factor in the survey. Higher scores indicate a higher frequency of specific sensory responses.
Vanderbilt Assessment Scale | 8 weeks
  Both parent and teacher assessment scales have two components: symptom assessment and impairment in performance. The symptom assessment component screens for symptoms relevant to inattentive and hyperactive ADHD subtypes. To meet criteria for ADHD diagnoses, one must have 6 positive responses to either the core 9 inattentive symptoms or core 9 hyperactive symptoms, or both.
  A positive response is either a score of 2 or 3 ("often" to "very often"). The final 8 questions of both versions ask the respondent to rate the child's performance in school and his or her interactions with others on a 1-5 scale, with 1-2 meaning "above average", 3 meaning "average", and 4-5 meaning "problematic".
  To meet the criteria for ADHD, there must be at least one score for the performance set that is a 5, or two scores that are at least 4, as these scores indicate impairment in performance.

CONTACTS AND LOCATIONS:
Overall Officials: Evren ERİK, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tse CYA, Lee HP, Chan KSK, Edgar VB, Wilkinson-Smith A, Lai WHE. Examining the impact of physical activity on sleep quality and executive functions in children with autism spectrum disorder: A randomized controlled trial. Autism. 2019 Oct;23(7):1699-1710. doi: 10.1177/1362361318823910. Epub 2019 Jan 20. PMID 30663324
- [Background] Xiao N, Shinwari K, Kiselev S, Huang X, Li B, Qi J. Effects of Equine-Assisted Activities and Therapies for Individuals with Autism Spectrum Disorder: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2023 Feb 1;20(3):2630. doi: 10.3390/ijerph20032630. PMID 36767996
- [Background] Kashefimehr B, Kayihan H, Huri M. The Effect of Sensory Integration Therapy on Occupational Performance in Children With Autism. OTJR (Thorofare N J). 2018 Apr;38(2):75-83. doi: 10.1177/1539449217743456. Epub 2017 Dec 27. PMID 29281930
- [Background] Padmanabha H, Singhi P, Sahu JK, Malhi P. Home-based Sensory Interventions in Children with Autism Spectrum Disorder: A Randomized Controlled Trial. Indian J Pediatr. 2019 Jan;86(1):18-25. doi: 10.1007/s12098-018-2747-4. Epub 2018 Jul 25. PMID 30043192
- [Background] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460